CLINICAL TRIAL: NCT05857917
Title: Virtual Reality for for Pain and Anxiety Distraction Strategy on Peritoneal Catheter Insertion: A Pilot Study
Brief Title: Virtual Reality for for Pain and Anxiety Distraction Strategy on Peritoneal Catheter Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wei Chen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITT-2023-130
Record Dates: First submitted 2023-04-19; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Renal Function Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Participants randomized into this group will be introduced to VR use and watch a VR video that introduces the operating room environment 1 day before surgery and play a soothing video through VR during the surgery.
  Interventions: Device: Virtual Reality
- Standard care group (No Intervention): The participants randomized to this group will receive the usual standard preoperative and intraoperative management.

INTERVENTIONS:
Device: Virtual Reality — Virtual reality in PD catheter insertion surgery in the pre- and intraoperative setting.
  Arms: VR group

SUMMARY:
This clinical trial aims to investigate the effect of VR application on reducing preoperative anxiety and the intraoperative and postoperative pain of patients who undergo peritoneal dialysis catheter insertion. The main questions it aims to answer are: 1) Whether preoperative VR application can reduce preoperative anxiety in patients undergoing peritoneal dialysis catheter insertion; 2) Whether intraoperative VR application can reduce intraoperative and postoperative pain in patients undergoing peritoneal dialysis catheter insertion; 3) Whether VR application can improve patients satisfaction of the operation. Participants will be randomly assigned to the VR group and control group, and participants in the VR group will be introduced to VR use and watch a VR video about the operating room environment 1 day before the surgery. During the procedure, participants in the VR group will watch a soothing video through the VR device. In contrast, participants in the control group will receive the usual preoperative and surgical procedures. Preoperative anxiety, intraoperative and postoperative pain, and patient satisfaction will be compared between the two arms.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is an important alternative treatment modality for end-stage renal disease. Patients are required to undergo catheter insertion prior to PD. However, Patients undergoing catheterization for the first time often experience preoperative anxiety, and the procedure is usually performed under local anesthesia. Moreover, patients under local anesthesia are prone to significant intraoperative pain and poor surgical cooperation, which compromises the procedure and leads to low patient satisfaction. In recent years, virtual reality (VR) has been found to reduce preoperative anxiety and acute or chronic pain in medical fields such as pediatrics and dentistry. It is a non-invasive, accessible, safe, and effective modality. There is a lack of research on the use of virtual reality technology in peritoneal dialysis catheterization, so this study proposes to study the effect of VR application on reducing preoperative anxiety and intraoperative and postoperative pain in patients using VR before and during catheter insertion.

The study is a prospective, randomized, controlled, single-center study. Patients who meet the enrollment criteria will be randomly assigned to either the VR group or the control group. The VR group will be introduced to the use of VR and watch a VR video introducing the operating room environment 1 day prior to surgery, and play soothing audio/video via VR during surgery; the control group will undergo routine preoperative and surgical procedures. Preoperative anxiety, intraoperative and postoperative pain, and patient satisfaction will be assessed between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, male or female.
* Patients receiving PD catheter insertion for the first time.
* Signed informed consent form.

Exclusion Criteria:

* Hearing and vision impairments, or affective disorder.
* Communication is not possible due to impaired cognitive ability.
* History of epilepsy or seizure.
* History of long-term use of pain medication (opioids).
* History of severe cardiac failure (NYHA IV), acute myocardial infarction, or severe acute infection in recent three months.
* Patients who refuse to use VR.
* Other conditions deemed unsuitable by physicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Procedure-related pain | recorded within 30 minutes after surgery
  Measured by Visual Analogue Scale (VAS) pain measurement scale divided from 0 to 10 where 0 is no pain and 10 worst pain that can be imagined.
Anxiety assessment 30 minutes before surgery | 30 minutes before surgery
  State-Trait Anxiety Scale (STAI) was applied in the preoperative period, and only the 20-item state scale construct was used.
Patient satisfaction | within 30 minutes after surgery
  5-point Likert verbal rating scale: 5, extremely satisfied; 4, satisfied; 3, undecided; 2, dissatisfied; 1, extremely dissatisfied.

SECONDARY OUTCOMES:
Postoperative analgesics usage | after the operation until discharge from hospital
  The use of paracetamol, NSAIDs, opioids, and other analgesics administered to the patients after surgery to relieve the pain caused by the operation.
Distribution of systolic blood pressure of patients in the intraoperative period | Baseline values are measured 30 minutes before the procedure, then the values at 5 minutes after the start of the procedure and every 15 minutes thereafter are recorded.
  Difference between the highest value during the operation and the baseline value.
Distribution of diastolic blood pressure of patients in the intraoperative period | Baseline values are measured 30 minutes before the procedure, then the values at 5 minutes after the start of the procedure and every 15 minutes thereafter are recorded.
  Difference between the highest value during the operation and the baseline value.
Distribution of pulse rates of patients in the intraoperative period | Baseline values are measured 30 minutes before the procedure, then the values at 5 minutes after the start of the procedure and every 15 minutes thereafter are recorded.
  Difference between the highest value during the operation and the baseline value.
Distribution of respiratory rates of patients in the intraoperative period | Baseline values are measured 30 minutes before the procedure, then the values at 5 minutes after the start of the procedure and every 15 minutes thereafter are recorded.
  Difference between the highest value during the operation and the baseline value.
Patient reported pain post procedure | recorded at 4 hours post operation, and 24 hour intervals to four days post operation.
  Measured by Visual Analogue Scale (VAS) pain measurement scale divided from 0 to 10 where 0 is no pain and 10 worst pain that can be imagined.

OTHER OUTCOMES:
VR Questionnaire | within 30 minutes after surgery
  Tolerability, feasibility and satisfaction of VR use
Catheter insertion related complications | through study completion, an average of 10 days
  including peri-operative complications (bleeding, bowel injury), mechanical complication (drainage failure, displacement, fluid leak), infective complications (exit site, tunnel, peritonitis), and other catheter insertion related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China